CLINICAL TRIAL: NCT01947556
Title: The Effect of Rapid-acting Insulin Injected by Needle-free Jet-injection in the Management of Hyperglycemia in Patients With Diabetes
Brief Title: Insulin by Jet-injection for Hyperglycemia in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, HM de Wit, MD, University Medical Center Nijmegen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PKPD_INSJ_3
Record Dates: First submitted 2013-09-02; First posted 2013-09-20 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; insulin administration; hyperglycaemia; insulin aspart
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insujet is tested first (Other): first procedure: experiment with the investigational product (Insujet pen)containing insulin aspart; second procedure: control device (conventional Novopen III insulin pen) contains insulin aspart.
  Interventions: Drug: insulin aspart
- insujet is tested second (Other): first procedure: experiment with the conventional Novopen III insulin pen containing insulin aspart; second procedure: investigational device (Insujet) contains insulin aspart.
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — After hyperglycaemia (18-23 mmol/l) has been reached (by decreasing or interrupting exogenous insulin administration 12-24 hours before the experiment), aspart insulin (in a dose of 1.5 times the amount of insulin needed to reduce blood glucose to 6 mmol/l calculated by the insulin-sensitivity factor) will be administered subcutaneously by Insujet pen or conventional insulin pen, on two separate occasions, or vice versa. The injection will be given by the subject under supervision of the research staff.
  Other Names: Novorapid

SUMMARY:
The purpose of this study is to compare the pharmacokinetic and pharmacodynamic profile of the rapid-acting insulin analogue aspart (Novorapid®) injected subcutaneously by jet-injection to that of the same insulin injected with a conventional pen in the management of hyperglycemia in subjects with diabetes

DETAILED DESCRIPTION:
Recently, we showed in both healthy, non-diabetic volunteers and in patients with type 1 (T1DM) and insulin-treated type 2 diabetes (T2DM) a 40-50% faster absorption of rapid-acting insulin analogues when administered by jet injection technology rather than by conventional insulin pen. The faster insulin action of insulin administration by jet injection may be especially advantageous for correction of hyperglycemia.

To investigate this, a open-label randomised controlled cross-over study will be performed in 20 adult patients (18-75 years) with T1DM or T2DM on basal-bolus insulin treatment.

The pharmacokinetic and pharmacodynamic profile of insulin aspart will be derived from the time-action profiles of insulin and glucose, respectively, in response to insulin (in a dose of 1.5 times the amount of insulin needed to reduce blood glucose to 6 mmol/l calculated by the insulin-sensitivity factor) after reaching hyperglycemia (18-23 mmol/l). All patients will be investigated twice, where on one occasion the jet-injector device will be used to inject insulin, and on the other occasion insulin will be injected with a conventional insulin pen. The order of these occasions will be randomised. Both devices will be operated by the patient after sufficient training. Ease of use will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 1 or 2
* Age 18-75 years
* Body-Mass Index ≥25 kg/m2 and ≤40 kg/m2
* Stable glycaemic control with HbA1c ≥48 (6.5%) and ≤86 mmol/mol (10%)
* Insulin treatment according to basal-bolus regimen, i.e. by multiple daily injections at least four times daily, or by subcutaneous insulin pump, for at least 12 months, use of metformin allowed

Exclusion Criteria:

* Inability to provide informed consent
* Insulin requirement of <34 or >200 units per day
* Treatment with systemic corticosteroids, immunosuppressive or cytostatic drugs
* Known allergy to aspart insulin
* Use of oral antidiabetic drugs other than metformin
* Symptomatic diabetic neuropathy
* History of a major cardiovascular disease event (myocardial infarction, stroke, symptomatic peripheral artery disease, coronary bypass surgery, percutaneous coronary or peripheral artery angioplasty) in the previous 6 months
* Pregnancy or the intention to become pregnant
* Renal disease (creatinine >150 μmol/l or MDRD-GFR <30 ml/min/1.73m2)
* Liver disease (aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range)
* Presence of any other medical condition that might interfere with the study protocol
* anemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
T-BG≥10 | participants will be followed for the duration of the study, an expected average of 4 weeks
  the time in minutes until plasma glucose concentration has dropped with ≥ 10mmol/l (T-BG≥10).

SECONDARY OUTCOMES:
T-BG5 and 8 (min) | participants will be followed for the duration of the study, an expected average of 4 weeks
  the time in minutes until plasma glucose values drop below 8 an 5 mmol/l, respectively
Rfall | participants will be followed for the duration of the study, an expected average of 4 weeks
  the slope of the glucose fall (mmol • l-1 • min-1), calculated from the time- glucose curve
BG-AUC 0-2h | participants will be followed for the duration of the study, an expected average of 4 weeks
  the area under the time-glucose curve, reflecting post-injection hyperglycaemic burden, from 0 to 2h after insulin injection.
BG-AUC 0-6h | participants will be followed for the duration of the study, an expected average of 4 weeks
  the area under the time-glucose curve (mmol • min-1 • l-1), from 0 to 6h after insulin injection.
C-INSmax (pmol/l) | participants will be followed for the duration of the study, an expected average of 4 weeks
  maximal insulin concentration
T-INSmax | participants will be followed for the duration of the study, an expected average of 4 weeks
  time to maximal insulin concentration in minutes(C-INSmax)
T-INSBL | participants will be followed for the duration of the study, an expected average of 4 weeks
  the time until plasma insulin values drop below baseline values (minutes)
INSAUC | participants will be followed for the duration of the study, an expected average of 4 weeks
  area under the insulin concentration curve (pmol • min-1 • l-1)(from timepoint 0), reflects total insulin absorption
T-INSAUC50% | participants will be followed for the duration of the study, an expected average of 4 weeks
  time until 50% of insulin absorption in minutes(mean residence time, MRT)

OTHER OUTCOMES:
NRS pain | participants will be followed for the duration of the study, an expected average of 4 weeks
  The amount of discomfort or pain and the ease of use experienced with the two administration methods using a numeric rating scale from 0 to 10 (will be administered 30 minutes after insulin administration)
hypoglycaemia | participants will be followed for the duration of the study, an expected average of 4 weeks
  Number of patients requiring exogenous glucose infusion to prevent hypoglycaemia (blood glucose ≤3.9 mmol/l) after insulin injection;
exogenous glucose | participants will be followed for the duration of the study, an expected average of 4 weeks
  Amount of exogenous glucose required to prevent hypoglycaemia after insulin injection
time exogenous glucose requirement | participants will be followed for the duration of the study, an expected average of 4 weeks
  Duration of time that exogenous glucose is required to prevent hypoglycaemia after insulin injection.

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan de Galan, MD PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands